CLINICAL TRIAL: NCT03565068
Title: A Multiple-dose Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and QTc Effect of MK-8189 in Participants With Schizophrenia and Healthy Participants.
Brief Title: A Safety, Tolerability, and Pharmacokinetics Study of MK-8189 in Participants With Schizophrenia and in Healthy Participants (MK-8189-007)
Acronym: MDCS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8189-007; MK-8189-007 (Other: Merck)
Record Dates: First submitted 2018-06-01; First posted 2018-06-21 (Actual); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — MK-8189

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Panel A (Healthy Participants): MK-8189 Monotherapy 4-24 mg (Experimental): Healthy participants will receive MK-8189 monotherapy orally once daily (QD) in escalating doses from 4 mg to 24 mg, as follows: Days 1-3: 4 mg, Days 4-6: 8 mg, Days 7-9: 12 mg, Days 10-12: 16 mg, Days 13-15: 20 mg, Days 16-18: 24 mg, depending on safety and tolerability.
  Interventions: Drug: MK-8189
- Panel A (Healthy Participants): Placebo Monotherapy (Placebo Comparator): Healthy participants will receive MK-8189 monotherapy matching placebo orally QD on Days 1-18.
  Interventions: Drug: Placebo
- Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4-24 mg (Experimental): Participants with Schizophrenia will receive MK-8189 monotherapy orally QD in escalating doses from 4 mg to 24 mg, as follows: Days 1-3: 4 mg, Days 4-6: 8 mg, Days 7-9: 12 mg, Days 10-12: 16 mg, Days 13-15: 20 mg, Days 16-18: 24 mg, depending on safety and tolerability.
  Interventions: Drug: MK-8189
- Panel B (Schizophrenia Participants): Placebo Monotherapy (Placebo Comparator): Participants with Schizophrenia will receive MK-8189 monotherapy matching placebo orally QD on Days 1-18.
  Interventions: Drug: Placebo
- Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4-24 mg (Experimental): In addition to background atypical antipsychotic (AAP) treatment, participants with Schizophrenia will receive MK-8189 add-on therapy orally QD in escalating doses from 4 mg to 24 mg, as follows: Days 1-3: 4 mg, Days 4-6: 8 mg, Days 7-9: 12 mg, Days 10-12: 16 mg, Days 13-15: 20 mg, Days 16-18: 24 mg, depending on safety and tolerability.
  Interventions: Drug: MK-8189; Drug: Background AAP Therapy
- Panel C (Schizophrenia Participants): Placebo Add-on Therapy (Placebo Comparator): In addition to background AAP treatment, participants with Schizophrenia will receive MK-8189 add-on therapy matching placebo orally QD on Days 1-18.
  Interventions: Drug: Placebo; Drug: Background AAP Therapy
- Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8-48 mg (Experimental): Participants with Schizophrenia will receive MK-8189 monotherapy orally QD in escalating doses from 8 mg to 48 mg, as follows: Days 1-3: 8 mg, Days 4-6: 16 mg, Days 7-9: 24 mg, Days 10-12: 36 mg, Days 13-15: 48 mg, depending on safety and tolerability.
  Interventions: Drug: MK-8189
- Panel D (Schizophrenia Participants): Placebo Monotherapy (Placebo Comparator): Participants with Schizophrenia will receive MK-8189 monotherapy matching placebo orally QD on Days 1-15.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8189 — MK-8189 4 mg tablet(s) will be administered orally QD for a total daily dose of 4 mg, 8 mg, 12 mg, 16 mg, 20 mg, 24 mg, 36 mg or 48 mg.
  Arms: Panel A (Healthy Participants): MK-8189 Monotherapy 4-24 mg; Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4-24 mg; Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4-24 mg; Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8-48 mg
Drug: Placebo — MK-8189 dose-matching placebo tablets will be administered orally QD.
  Arms: Panel A (Healthy Participants): Placebo Monotherapy; Panel B (Schizophrenia Participants): Placebo Monotherapy; Panel C (Schizophrenia Participants): Placebo Add-on Therapy; Panel D (Schizophrenia Participants): Placebo Monotherapy
Drug: Background AAP Therapy — Participants with schizophrenia in Panel C will be on background therapy with an AAP medication (e.g., olanzapine, quetiapine, paliperidone, asenapine, iloperidone, aripirprazole, lurasidone, risperidone [not to exceed daily dose of 6 mg], or ziprasidone) throughout the study. Participants should be on a stable and well tolerated treatment regimen for at least 2 months prior to screening. NOTE: clozapine is not allowed.
  Arms: Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4-24 mg; Panel C (Schizophrenia Participants): Placebo Add-on Therapy

SUMMARY:
This 4-panel study will evaluate the safety, tolerability, pharmacokinetics (PK) and corrected QT interval (QTc) effect of MK-8189 versus placebo, as monotherapy in healthy participants (Panel A) including those of Japanese descent, as monotherapy in participants with schizophrenia (Panel B), as add-on therapy in participants with schizophrenia (Panel C), and under an alternative dosing regimen as monotherapy in participants with schizophrenia (Panel D). Analysis of QTc effect will be exploratory. There will be no hypothesis testing in this study.

DETAILED DESCRIPTION:
As specified by Phase 1 protocol-flexible language in the protocol, modifications to the dose or dosing regimen can be made to achieve the scientific goals of the study objectives and/or to ensure appropriate safety of the study participants. The proposed doses for each Panel may be adjusted downward based on evaluation of observed safety, tolerability, and PK data.

ELIGIBILITY:
Inclusion Criteria

Panel A (Healthy Participants)

- If participant is of Japanese descent, both biological parents and all biological grandparents must be born in Japan.

Panels B and D (Participants with Schizophrenia; MK-8189 or Placebo Monotherapy / 15-Day Titration Monotherapy) - Is able to discontinue the use of all antipsychotic medication at least 5 days prior to the start of the treatment period and during the study period.

Panels B, C, and D (Participants with Schizophrenia; MK-8189 or Placebo Monotherapy / Add-on Therapy / 15-Day Titration Monotherapy)

* Meets diagnostic criteria for schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria with the onset of the first episode being no less than 2 years prior to screening and monotherapy with antipsychotics for treatment should be indicated.
* Is in the non-acute phase of their illness and clinically stable for 3 months prior to screening as demonstrated by: a.) no clinically significant change in dose of prescribed antipsychotic medication, or clinically significant change in antipsychotic medication to treat symptoms of schizophrenia for 2 months prior to screening; b.) no increase in level of psychiatric care due to worsening of symptoms of schizophrenia for 3 months prior to screening.
* Has a history of receiving and tolerating antipsychotic medication within the usual dose range employed for schizophrenia.
* Has a stable living situation in which the participant or a contact person can be reached by the investigator if there is a need for follow up.
* Participants with hypothyroidism, diabetes, high blood pressure, chronic respiratory conditions or other mild forms of these medical conditions could be considered as candidates for study enrollment if their condition is stable and the prescribed dose and regimen of medication is stable for at least 3 months prior to screening and there are no expected changes in co-medication during the study.
* Has regular bowel movements.

Panels A, B, C, and D

- A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

* Is not a woman of childbearing potential (WOCBP)
* Is a WOCBP and using a contraceptive method that is highly effective, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 14 days after the last dose of study intervention.

Exclusion Criteria

Panel A (Healthy Participants)

* Has a history of clinically diagnosed depression, anxiety disorder, or any history of psychiatric disorders having required drug treatment or hospitalization. Participants who have had situational depression more than 5 years before the start of the study may be enrolled in the study at the discretion of the investigator.
* Has a history of stroke, chronic seizures, or major neurological disorder.
* Has a history of dystonic reaction to antipsychotic, anti-emetic or related medication.
* Is at imminent risk of self-harm, based on clinical interview and responses on the Columbia Suicide Severity Rating Scale (C-SSRS), or of harm to others in the opinion of the investigator. Participants must be excluded if they report suicidal ideation with intent, with or without a plan or method (e.g., positive response to item 4 or 5 in assessment of suicidal ideation on the C-SSRS) in the past 5 years or suicidal behavior in their lifetime.
* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases. Participants with a remote history of uncomplicated medical events may be enrolled in the study at the discretion of the investigator.
* Is mentally or legally incapacitated, has a history of clinically significant psychiatric disorder of the last 5 years. Participants who have had situational depression may be enrolled in the study at the discretion of the investigator.
* Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies, beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study (including washout intervals between treatment periods), until the poststudy visit.
* Is a smoker and/or has used nicotine or nicotine-containing products (e.g., nicotine patch and electronic cigarette) within 3 months of screening.

Panels B, C, and D (Participants with Schizophrenia; MK-8189 or Placebo Monotherapy / Add-on Therapy / 15-Day Titration Monotherapy)

* Has evidence or history of a primary DSM-5 axis I psychiatric diagnosis other than schizophrenia or schizoaffective disorder per the allowed DSM-5 criteria within 1 month of screening.
* Has evidence or history of mental retardation, borderline personality disorder, anxiety disorder, or organic brain syndrome.
* Has a history of neuroleptic malignant syndrome or moderate to severe tardive dyskinesia (TD).
* Has a substance-induced psychotic disorder or behavioral disturbance thought to be due to substance abuse.
* Has a DSM-5 defined substance abuse or dependence disorder (excluding nicotine and caffeine) within three months of screening.
* Has a history of seizure disorder beyond childhood or is receiving treatment with any anticonvulsant to prevent seizures.
* Is at imminent risk of self-harm, based on clinical interview and responses on the C-SSRS, or of harm to others in the opinion of the investigator. Participants must be excluded if they report suicidal ideation with intent, with or without a plan or method (e.g., positive response to item 4 or 5 in assessment of suicidal ideation on the C-SSRS) in the past 2 months or suicidal behavior in the past 6 months.
* Has received treatment with clozapine for schizophrenia or treatment with monoamine oxidase inhibitors within 3 months of screening. For Panel C participants, has received a total daily dose of risperidone > 6 mg.
* Is unable to refrain from the use of co-medication with a moderate or strong inhibiting or inducing effect on cytochrome P450 (CYP) 3A (CYP3A) and/or CYP2C9 beginning approximately 2 weeks or 5 half- lives, whichever is longer, prior to administration of the initial dose of trial drug and throughout the trial or is unable to refrain from the use of sensitive substrates of CYP2B6. Unable to refrain from cyclic hormone replacement therapy. There may be certain medications that are permitted
* Has received a parenteral depot antipsychotic medication within 3 months of pre-trial (screening).

Panels A, B, C, and D

* Is a woman of childbearing potential (WOCBP) who has a positive serum pregnancy test at the screening visit or a positive urine pregnancy test within 48 hours before the first dose of study intervention. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has a history of cancer (malignancy). Exceptions include: (1) Participants with adequately treated nonmelanomatous skin carcinoma or carcinoma in situ of the cervix may participate in the study; (2) Participants with other malignancies which have been successfully treated ≥10 years prior to the prestudy (screening) visit where, in the judgment of both the investigator and treating physician, appropriate follow-up has revealed no evidence of recurrence from the time of treatment through the time of the prestudy (screening) visit (except those cancers identified at the beginning of this exclusion criteria); or (3) Participants, who, in the opinion of the study investigator, are highly unlikely to sustain a recurrence for the duration of the study.
* Has a clinically significant history or presence of sick sinus syndrome, first, second, or third degree atrioventricular (AV) block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QTc interval, or conduction abnormalities.
* Has history of repeated or frequent syncope, vasovagal episodes, or epileptic seizures.
* Has a family history of sudden death.
* Has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* Has a history of significant multiple and/or severe allergies (e.g., food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e., systemic allergic reaction) to prescription or non-prescription drugs or food.
* Has Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV) infection.
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to the prestudy (screening) visit. The window will be derived from the date of the last visit in the previous study.
* Has history or presence of risk factors for Torsade de Pointes (e.g., cardiac disease, heart failure, hypokalaemia or hypomagnesaemia, hypertrophy, cardiomyopathy, or family history of long QT syndrome). Plasma calcium must be within normal limits at screening and serum calcium must be within normal limits prior to dosing.
* Is under the age of legal consent.
* Has been in incarceration or imprisonment within 3 months prior to screening.
* Consumes greater than 3 glasses of alcoholic beverages per day. Participants who consume 4 glasses of alcoholic beverages per day may be enrolled at the discretion of the investigator.
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
* Is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 3 years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- California Clinical Trials ( Site 0001), Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol-specified dose modification, Panel C MK-8189 dose and schedule were modified, based on tolerability.
Groups:
- Panel A (Healthy Participants): MK-8189 Monotherapy 4-24 mg: Healthy participants received MK-8189 monotherapy orally once daily (QD) in escalating doses from 4 mg to 24 mg, as follows: Days 1-3: 4 mg, Days 4-6: 8 mg, Days 7-9: 12 mg, Days 10-12: 16 mg, Days 13-15: 20 mg, Days 16-18: 24 mg.
- Panel A (Healthy Participants): Placebo Monotherapy: Healthy participants received MK-8189 monotherapy matching placebo orally QD on Days 1-18.
- Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4-24 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD in escalating doses from 4 mg to 24 mg, as follows: Days 1-3: 4 mg, Days 4-6: 8 mg, Days 7-9: 12 mg, Days 10-12: 16 mg, Days 13-15: 20 mg, Days 16-18: 24 mg.
- Panel B (Schizophrenia Participants): Placebo Monotherapy: Participants with Schizophrenia received MK-8189 monotherapy matching placebo orally QD on Days 1-18.
- Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4-24 mg: In addition to background atypical antipsychotic (AAP) treatment, participants with Schizophrenia received MK-8189 add-on therapy orally QD in escalating doses from 4 mg to 24 mg, as follows: Days 1-3: 4 mg, Days 4-6: 8 mg, Days 7-9: 12 mg, Days 10-12: 16 mg, Days 13-15: 20 mg, Days 16-18: 24 mg.
- Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4-8 mg: In addition to background AAP treatment, participant with Schizophrenia received modified regimen of MK-8189 add-on therapy orally QD in escalating doses from 4 mg to 8 mg, as follows: Days 1-3: 4 mg, Days 4-11: 8 mg.
- Panel C (Schizophrenia Participants): Placebo Add-on Therapy: In addition to background AAP treatment, participants with Schizophrenia received MK-8189 add-on therapy matching placebo orally QD on Days 1-18.
- Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8-48 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD in escalating doses from 8 mg to 48 mg, as follows: Days 1-3: 8 mg, Days 4-6: 16 mg, Days 7-9: 24 mg, Days 10-12: 36 mg, Days 13-15: 48 mg.
- Panel D (Schizophrenia Participants): Placebo Monotherapy: Participants with Schizophrenia received MK-8189 monotherapy matching placebo orally QD on Days 1-15.
Period: Overall Study
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4-24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4-24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4-24 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4-8 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8-48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
Started | 12 | 4 | 12 | 4 | 12 | 1 | 4 | 17 | 9
Completed | 12 | 4 | 11 | 4 | 8 | 0 | 3 | 9 | 8
Not Completed | 0 | 0 | 1 | 0 | 4 | 1 | 1 | 8 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 5 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4-24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4-24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4-24 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4-8 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8-48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy | Total
Number analyzed (Participants) | 12 | 4 | 12 | 4 | 12 | 1 | 4 | 17 | 9 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (8.2) | 43.3 (15.4) | 49.3 (9.5) | 44.0 (8.9) | 44.3 (7.1) | 51.0 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed | 47.8 (7.2) | 44.4 (10.0) | 41.7 (9.6) | 43.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 6 | 0 | 5 | 1 | 2 | 8 | 4 | 36
  Male | 4 | 2 | 6 | 4 | 7 | 0 | 2 | 9 | 5 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 6
  Not Hispanic or Latino | 12 | 3 | 11 | 3 | 11 | 1 | 4 | 15 | 9 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 11 | 2 | 10 | 1 | 4 | 14 | 8 | 54
  White | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 10
  More than one race | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Area Under the Plasma-concentration Curve at Zero to 24 Hours Post-dose (AUC0-24hr) of MK-8189
Description: AUC was a measure of MK-8189 exposure assessed as a product of drug concentration and time, using a linear mixed effects model. To estimate AUC0-24hr per protocol blood samples were collected pre-dose, 2, 6, 8, 10, 12, 16, 24 hours post-dose for Panels A, B, C, D; no pre-dose samples collected on Day 18 (Panels A, B, C), Day 15 (Panel D). Samples were collected on Days 7, 10, 13, 16, 18 for Panels A, B; Days 9, 12, 15, 18 for Panel C; Days 1, 4, 7, 10, 13, 15 for Panel D. Per protocol AUC0-24hr was analyzed by panel, dose, dosing regimen; due to differing dosing regimen some arms/doses weren't applicable to some timepoints, shown by 0 participants analyzed in the table. Per dosing regimen the 4 mg, 8 mg (Panels A, B), 4 mg (Panel C) study arms weren't applicable to the protocol-specified timepoints/days of AUC0-24hr analysis and these arms were excluded. Geometric coefficient of variation (GCV) was reported as a percent. Per protocol placebo arms were excluded from AUC0-24hr analysis.
Time Frame: Pre-dose, 2, 6, 8, 10, 12, 16, 24 hours post-dose; no pre-dose on Day 18 (Panel A, B, C), Day 15 (Panel D); Panel A, B: Days 7, 10, 13, 16, 18; Panel C: Days 9, 12, 15, 18; Panel D: Days 1, 4, 7, 10, 13, 15
Population: All participants who got ≥1 dose of MK-8189, had AUC0-24hr data for Days 7, 10, 13, 16 or 18 (Panels A, B); Days 9, 12, 15 or 18 (Panel C); Days 1, 4, 7, 10, 13 or 15 (Panel D). Per protocol AUC0-24hr was analyzed by panel, dose, dosing regimen; based on dosing, some arms weren't applicable to some timepoints shown by 0 participants analyzed. The 4 mg, 8 mg (Panels A, B), 4 mg (Panel C) arms weren't applicable to the AUC0-24hr timepoints; per protocol these arms and placebo arms were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Groups:
- Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg: Healthy participants received MK-8189 monotherapy orally QD at a dose of 4 mg starting on Day 1 and continuing up to Day 3, based on participant tolerability
- Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg: Healthy participants received MK-8189 monotherapy orally QD at a dose of 8 mg starting on Day 4 and continuing up to Day 6, based on participant tolerability
- Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg: Healthy participants received MK-8189 monotherapy orally QD at a dose of 12 mg starting on Day 7 and continuing up to Day 9, based on participant tolerability
- Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg: Healthy participants received MK-8189 monotherapy orally QD at a dose of 16 mg starting on Day 10 and continuing up to Day 12, based on participant tolerability
- Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg: Healthy participants received MK-8189 monotherapy orally QD at a dose of 20 mg starting on Day 13 and continuing up to Day 15, based on participant tolerability
- Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg: Healthy participants received MK-8189 monotherapy orally QD at a dose of 24 mg starting on Day 16 and continuing up to Day 18, based on participant tolerability
- Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 4 mg starting on Day 1 and continuing up to Day 3, based on participant tolerability
- Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 8 mg starting on Day 4 and continuing up to Day 6, based on participant tolerability
- Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 12 mg starting on Day 7 and continuing up to Day 9, based on participant tolerability
- Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 16 mg starting on Day 10 and continuing up to Day 12, based on participant tolerability
- Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 20 mg starting on Day 13 and continuing up to Day 15, based on participant tolerability
- Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 24 mg starting on Day 16 and continuing up to Day 18, based on participant tolerability
- Panel B (Schizophrenia Participants): Placebo Monotherapy: Participants with Schizophrenia received MK-8189 monotherapy matching placebo orally QD from Days 1-18.
- Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg: In addition to background AAP treatment, participants with Schizophrenia received MK-8189 add-on therapy orally QD at a dose of 4 mg starting on Day 1 and continuing up to Day 3, based on participant tolerability
- Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg: In addition to background AAP treatment, participant with Schizophrenia received MK-8189 add-on therapy orally QD at a dose of 8 mg starting on Day 4 and continuing up to Day 11, based on participant tolerability
- Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg: In addition to background AAP treatment, participants with Schizophrenia received MK-8189 add-on therapy orally QD at a dose of 12 mg starting on Day 7 and continuing up to Day 9, based on participant tolerability
- Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg: In addition to background AAP treatment, participants with Schizophrenia received MK-8189 add-on therapy orally QD at a dose of 16 mg starting on Day 10 and continuing up to Day 12, based on participant tolerability
- Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg: In addition to background AAP treatment, participants with Schizophrenia received MK-8189 add-on therapy orally QD at a dose of 20 mg starting on Day 13 and continuing up to Day 15, based on participant tolerability
- Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg: In addition to background AAP treatment, participants with Schizophrenia received MK-8189 add-on therapy orally QD at a dose of 24 mg starting on Day 16 and continuing up to Day 18, based on participant tolerability
- Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 8 mg starting on Day 1 and continuing up to Day 3, based on participant tolerability
- Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 16 mg starting on Day 4 and continuing up to Day 6, based on participant tolerability
- Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 24 mg starting on Day 7 and continuing up to Day 9, based on participant tolerability
- Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 36 mg starting on Day 10 and continuing up to Day 12, based on participant tolerability
- Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg: Participants with Schizophrenia received MK-8189 monotherapy orally QD at a dose of 48 mg starting on Day 13 and continuing up to Day 15, based on participant tolerability
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
Number analyzed (Participants) | 0 | 0 | 11 | 11 | 10 | 10 | 0 | 0 | 0 | 11 | 11 | 10 | 10 | 0 | 0 | 1 | 10 | 8 | 7 | 7 | 0 | 17 | 16 | 15 | 13 | 11 | 0
nM*hr
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0
  Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 4640 (40.5) |  |  |  |  |
  Day 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0
  Day 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 10900 (72.1) |  |  |  |
  Day 7: number analyzed (Participants) | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0
  Day 7 |  |  | 8360 (42.5) |  |  |  |  |  |  | 11700 (32.9) |  |  |  |  |  |  |  |  |  |  |  |  |  | 14100 (106.6) |  |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 9 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 11400 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed | 11300 (47.9) |  |  |  |  |  |  |  |  |  |
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0
  Day 10 |  |  |  | 10200 (49.0) |  |  |  |  |  |  | 17200 (41.9) |  |  |  |  |  |  |  |  |  |  |  |  |  | 25100 (54.6) |  |
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 12 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 13800 (28.2) |  |  |  |  |  |  |  |  |
  Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Day 13 |  |  |  |  | 12200 (48.5) |  |  |  |  |  |  | 20200 (44.7) |  |  |  |  |  |  |  |  |  |  |  |  |  | 31800 (54.5) |
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 15700 (33.4) |  |  |  |  |  |  | 34400 (66.5) |
  Day 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 16 |  |  |  |  |  | 15600 (36.1) |  |  |  |  |  |  | 24600 (36.6) |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 18 |  |  |  |  |  | 13600 (59.6) |  |  |  |  |  |  | 26600 (38.3) |  |  |  |  |  |  | 18900 (30.8) |  |  |  |  |  |  |

2. Primary Outcome: The Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Per protocol, safety was analyzed by panel and dose. The number of participants who experienced one or more AEs was reported.
Time Frame: Up to ~32 days
Population: All participants who got ≥1 dose of study drug. Per protocol, safety was analyzed by panel and dose.
Measure: Count of Participants; unit: Participants
Groups:
- Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg: In addition to background AAP treatment, participants with Schizophrenia received MK-8189 add-on therapy orally QD at a dose of 8 mg starting on Day 4 and continuing up to Day 11, based on participant tolerability
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
Number analyzed (Participants) | 12 | 12 | 11 | 11 | 10 | 10 | 4 | 12 | 11 | 11 | 11 | 10 | 10 | 4 | 13 | 11 | 10 | 8 | 7 | 7 | 4 | 17 | 16 | 15 | 13 | 11 | 9
Participants | 5 | 3 | 4 | 5 | 2 | 5 | 3 | 4 | 3 | 4 | 8 | 5 | 7 | 4 | 6 | 8 | 5 | 5 | 4 | 4 | 1 | 8 | 8 | 5 | 5 | 8 | 9

3. Primary Outcome: The Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Per protocol, safety was analyzed by panel and dose. The number of participants who discontinued study treatment due to an AE was reported.
Time Frame: Up to ~18 days
Population: All participants who got ≥1 dose of study drug. Per protocol, safety was analyzed by panel and dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
Number analyzed (Participants) | 12 | 12 | 11 | 11 | 10 | 10 | 4 | 12 | 11 | 11 | 11 | 10 | 10 | 4 | 13 | 11 | 10 | 8 | 7 | 7 | 4 | 17 | 16 | 15 | 13 | 11 | 9
Participants | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 2

4. Secondary Outcome: Maximum Observed Post-dose Plasma Concentration (Cmax) of MK-8189
Description: Cmax was the maximum concentration of MK-8189 observed in plasma, assessed using a linear mixed effects model. To estimate Cmax, per protocol blood samples were collected pre-dose, 2, 6, 8, 10, 12, 16, 24 hours post-dose for Panels A, B, C, D; no pre-dose samples collected on Day 18 (Panels A, B, C), Day 15 (Panel D); additional post-dose samples collected at 36, 48 hours on Days 18 and 15. Samples were collected on Days 7, 10, 13, 16, 18 for Panels A, B; Days 9, 12, 15, 18 for Panel C; Days 1, 4, 7, 10, 13, 15 for Panel D. Per protocol Cmax was analyzed by panel, dose, dosing regimen; due to differing dosing regimen some arms/doses weren't applicable to some timepoints, shown by 0 participants analyzed in the table. Per dosing regimen, the 4 mg, 8 mg (Panels A, B), 4 mg (Panel C) study arms weren't applicable to the protocol-specified timepoints/days of Cmax analysis and were excluded. GCV was reported as a percent. Per protocol placebo arms were excluded from Cmax analysis.
Time Frame: Pre-dose, 2, 6, 8, 10, 12, 16, 24 hours post-dose; no pre-dose on Day 18 (Panel A, B, C), Day 15 (Panel D);additional 36, 48 hours post-dose on Days 18, 15; Panel A, B: Days 7, 10, 13, 16, 18; Panel C: Days 9, 12, 15, 18; Panel D:Days 1, 4, 7, 10, 13, 15
Population: All participants who got ≥1 dose of MK-8189, had Cmax data for Days 7, 10, 13, 16 or 18 (Panels A, B); Days 9, 12, 15 or 18 (Panel C); Days 1, 4, 7, 10, 13 or 15 (Panel D). Per protocol Cmax was analyzed by panel, dose, dosing regimen; based on dosing, some arms weren't applicable to some timepoints shown by 0 participants analyzed. The 4 mg, 8 mg (Panels A, B), 4 mg (Panel C) arms weren't applicable to the Cmax timepoints; per protocol these arms and placebo arms were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
Number analyzed (Participants) | 0 | 0 | 11 | 11 | 10 | 10 | 0 | 0 | 0 | 11 | 11 | 10 | 10 | 0 | 0 | 1 | 10 | 8 | 7 | 7 | 0 | 17 | 16 | 15 | 13 | 11 | 0
nM
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0
  Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 328 (42.8) |  |  |  |  |
  Day 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0
  Day 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 619 (52.5) |  |  |  |
  Day 7: number analyzed (Participants) | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0
  Day 7 |  |  | 481 (41.6) |  |  |  |  |  |  | 588 (33.7) |  |  |  |  |  |  |  |  |  |  |  |  |  | 920 (54.5) |  |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 9 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 591 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed | 566 (46.3) |  |  |  |  |  |  |  |  |  |
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0
  Day 10 |  |  |  | 613 (37.2) |  |  |  |  |  |  | 868 (41.5) |  |  |  |  |  |  |  |  |  |  |  |  |  | 1390 (46.1) |  |
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 12 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 693 (24.6) |  |  |  |  |  |  |  |  |
  Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Day 13 |  |  |  |  | 709 (47.1) |  |  |  |  |  |  | 1010 (45.0) |  |  |  |  |  |  |  |  |  |  |  |  |  | 1670 (51.9) |
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 801 (27.3) |  |  |  |  |  |  | 1890 (52.9) |
  Day 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 16 |  |  |  |  |  | 807 (34.0) |  |  |  |  |  |  | 1250 (37.7) |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 18 |  |  |  |  |  | 741 (48.0) |  |  |  |  |  |  | 1300 (36.8) |  |  |  |  |  |  | 972 (23.4) |  |  |  |  |  |  |

5. Secondary Outcome: Plasma Concentration at 24 Hours Post-dose (C24hr) of MK-8189
Description: C24hr was the concentration of MK-8189 observed in plasma at the 24-hour nominal sampling time after administration of MK-8189, assessed using a linear mixed effects model. To estimate C24hr, per protocol blood samples were collected 24 hours post-dose on Days 7, 10, 13, 16, 18 for Panels A, B; Days 9, 12, 15, 18 for Panel C; Days 1, 4, 7, 10, 13, 15 for Panel D. Per protocol C24hr was analyzed by panel, dose, dosing regimen; due to differing dosing regimen some arms/doses weren't applicable to some timepoints, shown by 0 participants analyzed in the table. Per dosing regimen, the 4 mg, 8 mg (Panels A, B), 4 mg (Panel C) study arms weren't applicable to the protocol-specified timepoints/days of C24hr analysis and were excluded. GCV was reported as a percent. Per protocol placebo arms were excluded from C24hr analysis.
Time Frame: 24 hours post-dose; Panel A, B: Days 7, 10, 13, 16, 18; Panel C: Days 9, 12, 15, 18; Panel D: Days 1, 4, 7, 10, 13, 15
Population: All participants who got ≥1 dose of MK-8189, had C24hr data for Days 7, 10, 13, 16 or 18 (Panels A, B); Days 9, 12, 15 or 18 (Panel C); Days 1, 4, 7, 10, 13 or 15 (Panel D). Per protocol C24hr was analyzed by panel, dose, dosing regimen; based on dosing, some arms weren't applicable to some timepoints shown by 0 participants analyzed. The 4 mg, 8 mg (Panels A, B), 4 mg (Panel C) arms weren't applicable to the C24hr timepoints; per protocol these arms and placebo arms were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
Number analyzed (Participants) | 0 | 0 | 11 | 6 | 10 | 10 | 0 | 0 | 0 | 11 | 11 | 10 | 10 | 0 | 0 | 1 | 10 | 8 | 6 | 7 | 0 | 17 | 16 | 14 | 13 | 11 | 0
nM
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0
  Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 287 (70.3) |  |  |  |  |
  Day 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0
  Day 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 480 (101.8) |  |  |  |
  Day 7: number analyzed (Participants) | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 0
  Day 7 |  |  | 310 (47.2) |  |  |  |  |  |  | 501 (37.9) |  |  |  |  |  |  |  |  |  |  |  |  |  | 567 (131.4) |  |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 9 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 416 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed | 490 (54.0) |  |  |  |  |  |  |  |  |  |
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0
  Day 10 |  |  |  | 392 (61.4) |  |  |  |  |  |  | 702 (46.9) |  |  |  |  |  |  |  |  |  |  |  |  |  | 890 (80.3) |  |
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 12 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 540 (39.1) |  |  |  |  |  |  |  |  |
  Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Day 13 |  |  |  |  | 418 (65.0) |  |  |  |  |  |  | 836 (57.0) |  |  |  |  |  |  |  |  |  |  |  |  |  | 1370 (47.5) |
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 651 (44.1) |  |  |  |  |  |  | 1160 (97.8) |
  Day 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 16 |  |  |  |  |  | 625 (39.7) |  |  |  |  |  |  | 949 (45.7) |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 18 |  |  |  |  |  | 433 (111.3) |  |  |  |  |  |  | 1010 (47.5) |  |  |  |  |  |  | 704 (39.0) |  |  |  |  |  |  |

6. Secondary Outcome: Time Post-dose to Maximum Observed Plasma Concentration (Tmax) of MK-8189
Description: Tmax was the actual sampling time at which maximum post-dose plasma concentration of MK-8189 was observed. To estimate Tmax, per protocol blood samples were collected pre-dose, 2, 6, 8, 10, 12, 16, 24 hours post-dose for Panels A, B, C, D; no pre-dose samples collected on Day 18 (Panels A, B, C), Day 15 (Panel D); additional post-dose samples collected at 36, 48 hours on Days 18 and 15. Samples were collected on Days 7, 10, 13, 16, 18 for Panels A, B; Days 9, 12, 15, 18 for Panel C; Days 1, 4, 7, 10, 13, 15 for Panel D. Per protocol Tmax was analyzed by panel, dose, dosing regimen; due to differing dosing regimen, some arms/doses weren't applicable to some timepoints, shown by 0 participants analyzed in the table. Per dosing regimen, the 4 mg, 8 mg (Panels A, B), 4 mg (Panel C) study arms weren't applicable to the protocol-specified timepoints/days of Tmax analysis and were excluded. Per protocol placebo arms were excluded from Tmax analysis.
Time Frame: as for outcome 4
Population: All participants who got ≥1 dose of MK-8189, had Tmax data for Days 7, 10, 13, 16 or 18 (Panels A, B); Days 9, 12, 15 or 18 (Panel C); Days 1, 4, 7, 10, 13 or 15 (Panel D). Per protocol Tmax was analyzed by panel, dose, dosing regimen; based on dosing, some arms weren't applicable to some timepoints shown by 0 participants analyzed. The 4 mg, 8 mg (Panels A, B), 4 mg (Panel C) arms weren't applicable to the Tmax timepoints; per protocol these arms and placebo arms were excluded.
Measure: Median (Full Range); unit: hr
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
Number analyzed (Participants) | 0 | 0 | 11 | 11 | 10 | 10 | 0 | 0 | 0 | 11 | 11 | 10 | 10 | 0 | 0 | 1 | 10 | 8 | 7 | 7 | 0 | 17 | 16 | 15 | 13 | 11 | 0
hr
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0
  Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 23.95 [12.00 to 24.00] |  |  |  |  |
  Day 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0
  Day 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 12.04 [0.00 to 23.98] |  |  |  |
  Day 7: number analyzed (Participants) | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0
  Day 7 |  |  | 12.02 [8.00 to 16.02] |  |  |  |  |  |  | 15.98 [6.00 to 23.95] |  |  |  |  |  |  |  |  |  |  |  |  |  | 16.03 [0.00 to 23.97] |  |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 9 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 12.00 [NA to NA] — Measure of dispersion could not be estimated due to low number of participants analyzed | 15.99 [2.00 to 23.92] |  |  |  |  |  |  |  |  |  |
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0
  Day 10 |  |  |  | 16.02 [10.03 to 23.95] |  |  |  |  |  |  | 16.07 [10.03 to 23.98] |  |  |  |  |  |  |  |  |  |  |  |  |  | 12.00 [0.00 to 23.95] |  |
  Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 12 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 11.09 [0.00 to 23.92] |  |  |  |  |  |  |  |  |
  Day 13: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Day 13 |  |  |  |  | 14.04 [0.00 to 16.10] |  |  |  |  |  |  | 16.05 [6.00 to 24.00] |  |  |  |  |  |  |  |  |  |  |  |  |  | 16.02 [8.00 to 16.15] |
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 16.00 [6.00 to 23.95] |  |  |  |  |  |  | 16.02 [6.05 to 16.13] |
  Day 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 16 |  |  |  |  |  | 13.99 [6.00 to 16.03] |  |  |  |  |  |  | 10.09 [6.00 to 23.93] |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 18 |  |  |  |  |  | 11.99 [8.00 to 16.03] |  |  |  |  |  |  | 12.05 [8.02 to 16.07] |  |  |  |  |  |  | 12.00 [6.00 to 16.07] |  |  |  |  |  |  |

7. Secondary Outcome: Apparent Total Plasma Clearance of MK-8189 (CL/F) on Day 18 (Panels A, B, C) and Day 15 (Panel D)
Description: CL/F was the apparent total clearance of MK-8189 in plasma over time, assessed as the rate at which MK-8189 was removed from the plasma. To estimate CL/F, per protocol blood samples were collected 2, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose on Day 18 for Panels A, B, C, and on Day 15 for Panel D. Per protocol CL/F was analyzed by panel, dose and dosing regimen. Due to differing dosing regimen, some arms/doses weren't applicable to some timepoints, shown by 0 participants analyzed in the table. Per dosing regimen, the 4 mg, 8 mg, 12 mg, 16 mg, 20 mg (Panels A, B, C), 8 mg, 16 mg, 24 mg, 36 mg (Panel D) study arms weren't applicable to the protocol-specified timepoints/days of CL/F analysis and were excluded. GCV was reported as a percent. Per protocol placebo arms were excluded from CL/F analysis.
Time Frame: 2, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose on Day 18 (Panel A, B, C) and Day 15 (Panel D)
Population: All participants who got ≥1 dose of MK-8189, had CL/F data for Day 18 (Panels A, B, C) or Day 15 (Panel D). Per protocol CL/F was analyzed by panel, dose, dosing regimen; based on dosing, some arms weren't applicable to some timepoints, shown by 0 participants analyzed. The 4 mg, 8 mg, 12 mg, 16 mg, 20 mg (Panels A, B, C), 8 mg, 16 mg, 24 mg, 36 mg (Panel D) arms weren't applicable to the CL/F timepoints; per protocol these arms and placebo arms were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hr
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 11 | 0
Liter/hr
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 3.65 (66.5) |
  Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 18 |  |  |  |  |  | 4.63 (59.6) |  |  |  |  |  |  | 2.36 (38.3) |  |  |  |  |  |  | 3.32 (30.8) |  |  |  |  |  |  |

8. Secondary Outcome: Apparent Volume of MK-8189 Distribution (Vd/F) on Day 18 (Panels A, B, C) and Day 15 (Panel D)
Description: Vd/F was the apparent volume of distribution of MK-8189 between the plasma and the rest of the body, after dose, assessed as the total volume of MK-8189 that would need to be uniformly distributed to achieve the desired plasma drug concentration. To estimate Vd/F, per protocol blood samples were collected 2, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose on Day 18 for Panels A, B, C, and on Day 15 for Panel D. Per protocol Vd/F was analyzed by panel, dose and dosing regimen. Due to differing dosing regimen, some arms/doses weren't applicable to some timepoints, shown by 0 participants analyzed in the table. Per dosing regimen, the 4 mg, 8 mg, 12 mg, 16 mg, 20 mg (Panels A, B, C), 8 mg, 16 mg, 24 mg, 36 mg (Panel D) study arms weren't applicable to the protocol-specified timepoints/days of Vd/F analysis and were excluded. GCV was reported as a percent. Per protocol placebo arms were excluded from Vd/F analysis.
Time Frame: 2, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose on Day 18 (Panel A, B, C) and Day 15 (Panel D)
Population: All participants who got ≥1 dose of MK-8189, had Vd/F data for Day 18 (Panels A, B, C) or Day 15 (Panel D). Per protocol Vd/F was analyzed by panel, dose, dosing regimen; based on dosing, some arms weren't applicable to some timepoints, shown by 0 participants analyzed. The 4 mg, 8 mg, 12 mg, 16 mg, 20 mg (Panels A, B, C), 8 mg, 16 mg, 24 mg, 36 mg (Panel D) arms weren't applicable to the Vd/F timepoints; per protocol these arms and placebo arms were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 10 | 0
Liter
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 47.1 (48.0) |
  Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 18 |  |  |  |  |  | 50.7 (48.6) |  |  |  |  |  |  | 37.2 (35.1) |  |  |  |  |  |  | 43.6 (39.1) |  |  |  |  |  |  |

9. Secondary Outcome: Time Required for Plasma Concentration of MK-8189 to Decrease by Half (Apparent Terminal Half-life [t1/2]) on Day 18 (Panels A, B, C) and Day 15 (Panel D)
Description: t1/2 was the time required to divide the plasma concentration of MK-8189 by half after reaching pseudo-equilibrium. At least three quantifiable terminal phase concentrations collected were used to calculate t1/2. To estimate t1/2, per protocol blood samples were collected 2, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose on Day 18 for Panels A, B, C, and on Day 15 for Panel D. Per protocol t1/2 was analyzed by panel, dose and dosing regimen. Due to differing dosing regimen, some arms/doses weren't applicable to some timepoints, shown by 0 participants analyzed in the table. Per dosing regimen, the 4 mg, 8 mg, 12 mg, 16 mg, 20 mg (Panels A, B, C), 8 mg, 16 mg, 24 mg, 36 mg (Panel D) study arms weren't applicable to the protocol-specified timepoints/days of t1/2 analysis and were excluded. GCV was reported as a percent. Per protocol placebo arms were excluded from t1/2 analysis.
Time Frame: 2, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose on Day 18 (Panel A, B, C) and Day 15 (Panel D)
Population: All participants who got ≥1 dose of MK-8189, had t1/2 data for Day 18 (Panels A, B, C) or Day 15 (Panel D). Per protocol t1/2 was analyzed by panel, dose, dosing regimen; based on dosing, some arms weren't applicable to some timepoints, shown by 0 participants analyzed. The 4 mg, 8 mg, 12 mg, 16 mg, 20 mg (Panels A, B, C), 8 mg, 16 mg, 24 mg, 36 mg (Panel D) arms weren't applicable to the t1/2 timepoints; per protocol these arms and placebo arms were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 10 | 0
hr
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 8.25 (20.0) |
  Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 18 |  |  |  |  |  | 7.60 (29.7) |  |  |  |  |  |  | 10.9 (25.5) |  |  |  |  |  |  | 9.10 (19.2) |  |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: Serious AEs, Non-serious AEs: Up to ~32 Days, All-cause mortality: Up to ~21 months
Description: Safety was analyzed by panel and by dose, in all participants who received at least one dose of the study drug.
Arm/Group | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg | Panel A (Healthy Participants): Placebo Monotherapy | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel B (Schizophrenia Participants): Placebo Monotherapy | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg | Panel C (Schizophrenia Participants): Placebo Add-on Therapy | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg | Panel D (Schizophrenia Participants): Placebo Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/11 | 0/10 | 0/10 | 0/4 | 0/12 | 0/11 | 0/11 | 0/11 | 0/10 | 0/10 | 0/4 | 0/13 | 0/11 | 0/10 | 0/8 | 0/7 | 0/7 | 0/4 | 0/17 | 0/16 | 0/15 | 0/13 | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/11 | 0/10 | 0/10 | 0/4 | 0/12 | 0/11 | 0/11 | 0/11 | 0/10 | 0/10 | 0/4 | 0/13 | 0/11 | 0/10 | 0/8 | 0/7 | 0/7 | 0/4 | 0/17 | 0/16 | 0/15 | 1/13 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 5/12 | 3/12 | 4/11 | 5/11 | 2/10 | 5/10 | 3/4 | 4/12 | 3/11 | 4/11 | 8/11 | 5/10 | 7/10 | 4/4 | 6/13 | 8/11 | 5/10 | 5/8 | 4/7 | 4/7 | 1/4 | 8/17 | 8/16 | 5/15 | 4/13 | 8/11 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg (N=12) | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg (N=12) | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg (N=11) | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg (N=11) | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg (N=10) | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg (N=10) | Panel A (Healthy Participants): Placebo Monotherapy (N=4) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg (N=12) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg (N=11) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg (N=11) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg (N=11) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg (N=10) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg (N=10) | Panel B (Schizophrenia Participants): Placebo Monotherapy (N=4) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg (N=13) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg (N=11) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg (N=10) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg (N=8) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg (N=7) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg (N=7) | Panel C (Schizophrenia Participants): Placebo Add-on Therapy (N=4) | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg (N=17) | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg (N=16) | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg (N=15) | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg (N=13) | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg (N=11) | Panel D (Schizophrenia Participants): Placebo Monotherapy (N=9)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A (Healthy Participants): MK-8189 Monotherapy 4 mg (N=12) | Panel A (Healthy Participants): MK-8189 Monotherapy 8 mg (N=12) | Panel A (Healthy Participants): MK-8189 Monotherapy 12 mg (N=11) | Panel A (Healthy Participants): MK-8189 Monotherapy 16 mg (N=11) | Panel A (Healthy Participants): MK-8189 Monotherapy 20 mg (N=10) | Panel A (Healthy Participants): MK-8189 Monotherapy 24 mg (N=10) | Panel A (Healthy Participants): Placebo Monotherapy (N=4) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 4 mg (N=12) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 8 mg (N=11) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 12 mg (N=11) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 16 mg (N=11) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 20 mg (N=10) | Panel B (Schizophrenia Participants): MK-8189 Monotherapy 24 mg (N=10) | Panel B (Schizophrenia Participants): Placebo Monotherapy (N=4) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 4 mg (N=13) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 8 mg (N=11) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 12 mg (N=10) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 16 mg (N=8) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 20 mg (N=7) | Panel C (Schizophrenia Participants): MK-8189 Add-on Therapy 24 mg (N=7) | Panel C (Schizophrenia Participants): Placebo Add-on Therapy (N=4) | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 8 mg (N=17) | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 16 mg (N=16) | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 24 mg (N=15) | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 36 mg (N=13) | Panel D (Schizophrenia Participants): MK-8189 Monotherapy 48 mg (N=11) | Panel D (Schizophrenia Participants): Placebo Monotherapy (N=9)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic heart rate response increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Dissociation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT03565068/Prot_SAP_000.pdf